CLINICAL TRIAL: NCT06814548
Title: Immune Checkpoint Inhibitors (ICIs) Retreatment in Second-line Treatment of Advanced Gastric Cancer: a Retrospective, Real-world Study
Status: Not yet recruiting | Type: Observational
Sponsor: Yongxu Jia (Other)
Responsible Party: Sponsor-Investigator, Yongxu Jia, Doctor, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Other Study IDs: GC-2L-ICI-2024
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer, Gastroesophageal Junction Cancer; Immune Checkpoint Inhibitors (ICIs); Second-line; Retreatment
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Immunohistochemical detection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ICIs retreatment: Histologically confirmed metastatic or advanced GC/GEJC; Received at least 2 cycles of anti-PD-1 or PD-L1 based therapy in the first-line setting; Receiving at least 2 cycles of ICI-based second-line therapy; ECOG PS 0 or 1; Radiographic response was also assessed during treatment and survival.
  Interventions: Other: ICIs(Immune checkpoint inhibitors)

INTERVENTIONS:
Other: ICIs(Immune checkpoint inhibitors) — N

SUMMARY:
This is a single-center, retrospective, observational, real-world study. We collected general and clinical data of patients with advanced gastric cancer who were admitted to the First Affiliated Hospital of Zhengzhou University from January 2018 to July 2024.

DETAILED DESCRIPTION:
All patients received combination therapy with ICIs inhibitors for at least 2 cycles in the first-line and at least 2 cycles of ICI inhibitor-based therapy in the second-line after first-line progression. The efficacy and safety of treatment were evaluated, including overall survival (OS), progression-free survival (PFS), objective response rate (ORR), disease control rate (DCR), Pattern of immune progression after cross-line therapy, grade 3-5 treatment-related adverse events (TRAEs), and immune-related adverse events (irAEs). Cox regression model was used to investigate the influence of multiple factors on survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or advanced GC/GEJC;
* Received at least 2 cycles of anti-PD-1 or PD-L1 based therapy in the first-line setting;
* Receiving at least 2 cycles of ICI-based second-line therapy;
* ECOG PS 0 or 1;
* Radiographic response was also assessed during treatment and survival.

Exclusion Criteria:

* patients had other malignancies within the past 5 years;
* lack of survival and clinical efficacy data;
* combined radiotherapy regimens in the second-line treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients received combination therapy with ICIs inhibitors for at least 2 cycles in the first-line and at least 2 cycles of ICI inhibitor-based therapy in the second-line after first-line progression.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 12 months
  Progression-free survival (PFS per RECIST 1.1) is defined as the time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first
overall survival (OS) | 12 months
  Progression-free survival (PFS per RECIST 1.1) is defined as the time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first

SECONDARY OUTCOMES:
objective response rate (ORR) | 12 months
  The proportion of subjects with complete response (CR) and partial response (PR) in total subjects
disease control rate (DCR) | 12 months
  The proportion of subjects with complete response (CR) and partial response (PR) and stable disease (SD) in total subjects
safety | 12 months
  Adverse events (AEs) were graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03.

IPD SHARING:
Plan to Share IPD: Yes